CLINICAL TRIAL: NCT04267627
Title: A Nurse-Led Telemedicine Videoconferencing Intervention to Improve Access to Supportive Cancer Survivorship Care for Rural Virginians
Brief Title: Telemedicine Nurse-Led Intervention for Rural Cancer Survivors
Acronym: CARING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Pamela DeGuzman, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20991
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Neoplasm; Survivorship
Keywords: Telemedicine; Cancer Survivorship; Rural Health Disparities
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nursing; Counseling

STUDY DESIGN:
Intervention Model Description: Three-arm trial evaluating CARING delivered over telemedicine vs. CARING delivered face-to-face vs. usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): No intervention.
- CARING with telemedicine (Experimental): Patients will receive the nurse-led supportive care intervention over telemedicine videoconferencing from home or from a satellite telemedicine site in Virginia.
  Interventions: Behavioral: Comprehensive Assistance: Rural Interventions, Nursing, and Guidance (CARING)
- CARING face-to-face (Experimental): Patients will receive the nurse-led supportive care intervention in person.
  Interventions: Behavioral: Comprehensive Assistance: Rural Interventions, Nursing, and Guidance (CARING)

INTERVENTIONS:
Behavioral: Comprehensive Assistance: Rural Interventions, Nursing, and Guidance (CARING) — Cancer-related distress will be assessed using the NCCN Distress Thermometer amended to include HNC-specific areas of distress. For those participants experiencing high rates of distress, the nurse will provide targeted distress education. Education for participants exhibiting successful distress self-management, or with distress that has already resolved will focus on reinforcing surveillance and health promotion information contained in the Survivorship Care Plan. When indicated, the nurse will discuss potential referrals to support services with the patient, and they will decide jointly which referrals will be beneficial. Following the visits, the nurse will make agreed upon referrals using existing cancer center pathways, documenting these in the medical record. The nurse will follow-up with the patient via telephone 6 weeks following the telemedicine visit to determine uptake of the referral, documenting all referral information in the electronic medical record.
  Arms: CARING face-to-face; CARING with telemedicine

SUMMARY:
This study will evaluate the impact, cost-effectiveness, and patient perspectives of Comprehensive Assistance: Rural Intervention, Nursing, and Guidance (CARING), a nurse-led supportive care protocol delivered using telemedicine videoconferencing aimed at reducing unmet needs in a rural head and neck cancer population. Specific aims: 1) Test the efficacy of CARING, delivered with and without telemedicine, compared to a control group. 2) Conduct a cost-effectiveness analysis of a nurse-led telemedicine visit. 3) Evaluate patient perceptions of a telemedicine intervention. Design: We will use a three-arm randomized control design to determine the efficacy of CARING delivered face-to-face, vs. CARING over telemedicine, vs. usual care. Costs will be determine for incremental cost effectiveness analysis, with quality of life years as the effectiveness variable. Patient perceptions will be evaluated qualitatively using the Practical, Robust Implementation and Sustainability Model (PRISM), designed to evaluate translation of research into practice and quantitatively using the Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ). Sample: We will enroll 450 head and neck cancer survivors of any stage who have completed treatment within the last 6 weeks (address over sampling of rural). Procedures: Following randomization, those in the intervention arm will either receive the nurse-led intervention in a clinic setting or over telemedicine videoconferencing 6 weeks following their in-person, end of treatment medical visit. Assessments at baseline, 6 weeks following the intervention, and 6 months following the intervention will document unmet needs using the Short Form Survivorship Unmet Needs (SF-SUNS) and quality of life using the Functional Assessment of Cancer Therapies- Head and Neck (FACT-HN) and the TSUQ and PRISM-guided questionnaires immediately following intervention. Health utilization costs at the societal and health system levels will be collected from the electronic medical record and patient interviews.

DETAILED DESCRIPTION:
Once cancer treatment has concluded (a phase called "extended survivorship") some cancer survivors continue to experience physical and psychosocial morbidities, and short-term and late effects of treatment, all of which can impact survivors' mental health, quality of life, and occupational and social functioning. Continued deficits in post-treatment health and function are termed survivorship unmet needs. Survivors of head and neck cancer (HNC; defined as cancer of the oral cavity, pharynx, larynx, sinuses, nasal cavity, and salivary glands) suffer numerous and often life-altering unmet needs including lingering pain, altered speech and eating, and facial disfigurement. Few interventions exist to connect HNC survivors with resources to address physical and psychosocial sequelae, and accordingly HNC survivors have high unmet needs. Rural survivors are even less likely to have their post-treatment needs met. The University of Virginia (UVa) Emily Couric Clinical Cancer Center (EC4) serves a largely rural catchment area where patients travel up to 6 hours to receive treatment. The EC4 offer a range of supportive care resources to assist HNC survivors during treatment, but once treatment is over, rural survivors are less likely to know of, let alone make use of these resources. Using resources of the well-established UVa Center for Telehealth (CFT) our intervention connects rural survivors with a nurse-led supportive care visit using telemedicine videoconferencing.

Preliminary data from Comprehensive Assistance: Rural Intervention, Nursing, and Guidance (CARING), a nurse-led, protocol-driven visit delivered over telemedicine videoconferencing suggests that supplementing medical follow-up with a face-to-face nursing visit over telemedicine works to overcome access barriers for rural survivors, and may reduce unmet needs, all without the need for the patient to travel to the EC4. Importantly, because of the extensive network and capabilities of the CFT we are able to offer the intervention either in patient's own home or through one of UVa's active telemedicine sites throughout the state. During the pilot intervention 35% (7/20) of participants were successfully referred to and connected with a supportive care provider. Pilot data suggests that a nurse-led proactive unmet needs intervention may overcome the stigma associated with asking for or accepting psychosocial help among rural residents, which can further complicate the provision of supportive care to this population.

Identifying the optimal approach to address rural survivors' unmet needs, we next need to determine if the nurse protocol or the telemedicine modality (or both) are driving intervention success. Health systems and policy makers considering adopting this model of care need understand to incremental costs and cost-effectiveness of providing a nurse-led protocol delivered via telemedicine. Rural and older populations may experience more difficulties adopting health technology; thus we need to determine patients' perspectives on the use and usefulness of the intervention.

Aim 1. Test the efficacy of CARING, delivered with and without telemedicine, compared to a control group. Hypothesis 1: HNC survivors who receive the CARING intervention will have a significantly larger reduction in unmet needs. Preliminary data revealed that HNC survivors of later cancer stage, longer distance to care, and receiving a home intervention, were more likely to accept a referral to address their unmet needs. We will determine the impact of those factors, as well as rurality, home broadband access, SES, race, ethnicity, and sex, on reduction in survivorship unmet needs. Hypothesis 2: Rural HNC survivors will be more likely to attend a home-based telemedicine intervention than an in-person visit. We will compare attendance rates of rural HNC survivors between those who receive a telemedicine home-based intervention and an in-person visit.

Aim 2. Conduct a cost-effectiveness analysis of a nurse-led telemedicine visit. We will calculate the ratio of incremental costs of delivering the intervention compared to the improvement in quality of life. Compare the relative costs of survivorship care delivered 1) with or without the CARING telemedicine intervention and 2) with or without the CARING intervention (without telemedicine) from both societal and health system perspectives. Analyze cost-effectiveness models for early and late stage cancers, and rural/non-rural survivors.

Aim 3. Evaluate patient perceptions of a telemedicine intervention. Hypothesis 3: Participants will report both the nurse interaction and minimizing travel as benefits of the intervention and technology use a barrier. Survey participants to determine intervention patient-centeredness, barriers, seamlessness of transition between program elements, access, and burden of participation in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Head and Neck Cancer
* Anticipated to be within 3 months of end of treatment
* At least 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number and type of Unmet Needs | baseline
  Survivorship Unmet Needs Survey- Short Form. 30 question scale with 0-4 rating for each item. Overall scores range 0-120. Lower scores indicated fewer unmet needs.
Number and type of Unmet Needs | 6 weeks post intervention
  Survivorship Unmet Needs Survey- Short Form. 30 question scale with 0-4 rating for each item. Overall scores range 0-120. Lower scores indicated fewer unmet needs.
Number and type of Unmet Needs | 6 monthspost intervention
  Survivorship Unmet Needs Survey- Short Form. 30 question scale with 0-4 rating for each item. Overall scores range 0-120. Lower scores indicated fewer unmet needs.
Quality of Life rating | baseline
  Functional Assessment of Cancer Therapies- Head and Neck (FACT-HN). Quality of life scale with 4 sub-scales and 12 items each related specifically to head and neck cancer quality of life. The Physical Health scale has 7 items, each rated 0-4. Scores range from 0-28 with a lower score indicating better quality of life. The Social Well Being scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The Emotional Well Being scale has 6 items, each rated 0-4. Scores range from 0-24 with a lower score indicating better quality of life. The Functional scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The remaining 12 items are all scored as 0-4 each, range for each item 0-4 with higher or lower score indicating better quality life depending on each individual item.
Quality of Life rating | 6 weeks post intervention
  Functional Assessment of Cancer Therapies- Head and Neck (FACT-HN). Quality of life scale with 4 sub-scales and 12 items each related specifically to head and neck cancer quality of life. The Physical Health scale has 7 items, each rated 0-4. Scores range from 0-28 with a lower score indicating better quality of life. The Social Well Being scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The Emotional Well Being scale has 6 items, each rated 0-4. Scores range from 0-24 with a lower score indicating better quality of life. The Functional scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The remaining 12 items are all scored as 0-4 each, range for each item 0-4 with higher or lower score indicating better quality life depending on each individual item.
Quality of Life rating | 6 months post intervention
  Functional Assessment of Cancer Therapies- Head and Neck (FACT-HN). Quality of life scale with 4 sub-scales and 12 items each related specifically to head and neck cancer quality of life. The Physical Health scale has 7 items, each rated 0-4. Scores range from 0-28 with a lower score indicating better quality of life. The Social Well Being scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The Emotional Well Being scale has 6 items, each rated 0-4. Scores range from 0-24 with a lower score indicating better quality of life. The Functional scale has 7 items, each rated 0-4. Scores range from 0-28 with a higher score indicating better quality of life. The remaining 12 items are all scored as 0-4 each, range for each item 0-4 with higher or lower score indicating better quality life depending on each individual item.

SECONDARY OUTCOMES:
telemedicine usefulness and satisfaction | within one week of intervention
  Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ). The TSUQ has 2 domains and a total of 21 items, the Video Visits domain (11 items) and the Use and Impact domain (10 items) each measured on a scale 1-5. The range of scores for Video Visits domain is 11-55 with a higher score indicating more satisfaction with video visits, and the Use and for the Use and Impact domain is 10-50, with higher scores indicating more usefulness to impact health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela B DeGuzman, PhD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No